CLINICAL TRIAL: NCT04085874
Title: Effectiveness of Optimized Food-Based Recommendations to Improve Dietary Practice, Intake of Problem Nutrient, Nutritional Status and Lipid Profile Among Minangkabau Women of Reproductive Age With Dyslipidemia
Brief Title: Effectiveness of Food-Based Recommendations for Minangkabau Women of Reproductive Age With Dyslipidemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Politeknik Kesehatan Kemenkes Padang (Other)
Collaborators: Indonesia University (Other)
Responsible Party: Principal Investigator, Gusnedi, Associate Professor, Politeknik Kesehatan Kemenkes Padang
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-12-1376
Record Dates: First submitted 2019-09-04; First posted 2019-09-11 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Dietary Habits; Nutrient Deficiency; Obesity; Dyslipidemias
Keywords: Nutrition intervention; Food-Based Recommendations; dietary practices; women of reproductive age; dyslipidemia
MeSH Terms: conditions — Feeding Behavior; Obesity; Dyslipidemias | interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FBR group (Experimental): weekly home visit and monthly group meeting for 12 weeks
  Interventions: Behavioral: Promotion of Food-based recommendations
- non-FBR group (Active Comparator): once nutrition counseling from standard health care services
  Interventions: Behavioral: Nutrition counseling from standard health services care

INTERVENTIONS:
Behavioral: Promotion of Food-based recommendations — Prolonged contact through weekly home visits and monthly group meeting for 12 weeks
  Other Names: Nutrition education
  Arms: FBR group
Behavioral: Nutrition counseling from standard health services care — once nutrition counselling from health services
  Other Names: Standard nutrition care
  Arms: non-FBR group

SUMMARY:
This study aimed to assess effectiveness of promoting the optimized Food-based recommendations (FBRs) for improving dietary practices, nutrient intakes, nutritional status and lipid profile among Minangkabau women of reproductive age with dyslipidemia in a community setting. A cluster randomized community-based trial was conducted in Padang City, West Sumatra, Indonesia. Subjects are Minagabau women of reproductive age (20-44 y) with dyslipidemia. The subjects were assigned either into FBR group (n=48) that involved in 12-weeks prolonged contact of FBRs promotion or into non-FBR group, that received once nutrition counselling from usual standard of nutrition program. Baseline and end-line lipid profiles, nutritional status, dietary practice and nutrient intake data were assessed through biochemical assessment, anthropometri, and interview structured questionaire.

DETAILED DESCRIPTION:
This study was conducted in two sequential phases. The first stage was a formative phase in the form of observational survey to develop and validate food-based recommendations (FBRs). The second phase was an intervention study to assess the effectiveness of the FBRs in improving dietary practice, the intake of problem nutrient, nutritional status and lipid profile of the subject.

Sample size for intervention per group (n=60/group; 2 groups) was expected to detect mean(±SD) differences in LDL-cholesterol concentration (as an secondary outcome) of 14±20 mg/dL as observed in a previous study in other area, with assumption of 80% power and 25% loss of follow up. Potential subjects were identified prior to dyslipidemia screening before intervention. Field nutritionist and volunteer cadres were requested to identify and list women of reproductive age fulfilling the inclusion criteria living in selected sites. An invitation letter was sent to all identified eligible subjects to visit appointed field laboratory to perform blood measurement. Inform consent was signed by all potential participants before blood measurement.

This study did not compare an intervention group (FBR group) with a true control group, but with a comparison group that received once nutrition counselling from usual nutrition health program (non-FBR group). Drawing on concepts of Plan Behavior Theory, persuasive FBR promotion was designed to influence subjects' attitude, subjective norms, perceive behavior control related to dyslipidemia and dietary management, and intention to change. Participants were prompted to set goals for themselves to improve their dietary practices in order to fulfill their nutrient requirements, improve nutritional status and lipid profile.

ELIGIBILITY:
Inclusion Criteria:

* women of reproductive age (20-44 years);
* native Minangkabau ethnic (both father and mother from the Minangkabau tribe);
* had abnormal one of isolated blood lipid profiles (cholesterol > 200 mg / dl, LDL-cholesterol >100 mg / dl, HDL < 60 mg/dl, TG > 150 mg/dl);
* signing a written inform consent.

Exclusion Criteria:

* in pregnancy;
* having a history or active smoker and alcoholic addict;
* has a history of heart disease, diabetes, asthma, cancer, chronic digestive tract disorders, hemophilia and other chronic diseases;
* routinely taking cholesterol-lowering or blood pressure medications;
* vegetarians;
* use estrogen therapy;
* are participating in other studies.

Ages: 20 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women of reproductive age
Enrollment: 123 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2019-05-05 (Actual); Study Completion 2019-06-10 (Actual)

PRIMARY OUTCOMES:
Change in Dietary practice | baseline (before the intervention) and end-line (after 12-weeks intervention)
  Change in food consumption from baseline at 12-week intervention, evaluated based on participant's compliance to the Optimized Food-Based Recommendations. The compliance were measured using one-week Food Frequency Questionnaire (FFQ), stated in servings/week for staple foods. snacks, animal protein (sea fish, eggs, poultry), soy protein (tofu/tempeh), potato, fruits,dark green vegetables (DGLV), total vegetables and fried foods. The recommendations (servings/week) for those food groups/items was 14-21, 7-14, minimum 5, 3-4, 2-3,minimum 7,minimum 5, minimum 7, minimum 5, minimum 14, and maximum 14 respectively. Those who complied with the recommendations was scored 1 for each recommendations, and 0 for those who did not. The total score for the compliance to the FBRs was 0-11. Higher score represents better participant's compliance
Change in energy intake | baseline (before intervention and end-line (after 12-weeks interventions)
  Change from baseline at 12-week intervention for energy intake( in Kcal). The intake was measured through interview using two replicates 24-hour food recall on non-consecutive days. The foods were converted to energy and nutrients based on Indonesia food composition tables available in nutrisurvey software
Change in protein intake | baseline (before intervention and end-line (after 12-weeks interventions)
  Change from baseline at 12-week intervention for protein intake( in gram). The intake was measured through interview using two replicates 24-hour food recall on non-consecutive days. The foods were converted to energy and nutrients based on Indonesia food composition tables available in nutrisurvey software
Change in total fat intake | baseline (before intervention and end-line (after 12-weeks interventions)
  Change from baseline at 12-week intervention for total fat intake( in gram). The intake was measured through interview using two replicates 24-hour food recall on non-consecutive days. The foods were converted to energy and nutrients based on Indonesia food composition tables available in nutrisurvey software.
Change in carbohydrate intake | baseline (before intervention and end-line (after 12-weeks interventions)
  Change from baseline at 12-week intervention for carbohydrate intake ( in gram)
Change in poly unsaturated fatty acids (PUFA) intake | baseline (before intervention and end-line (after 12-weeks interventions)
  Change from baseline at 12-week intervention for PUFA intake ( in gram). The intake was measured through interview using two replicates 24-hour food recall on non-consecutive days. The foods were converted to energy and nutrients based on Indonesia food composition tables available in nutrisurvey software.
Change in mono unsaturated fatty acids (MUFA) intakes | baseline (before intervention and end-line (after 12-weeks interventions)
  Change from baseline at 12-week intervention for MUFA intake ( in gram). The intake was measured through interview using two replicates 24-hour food recall on non-consecutive days. The foods were converted to energy and nutrients based on Indonesia food composition tables available in nutrisurvey software.
Change in saturated fatty acids (SFA) intakes | baseline (before intervention and end-line (after 12-weeks interventions)
  Change from baseline at 12-week intervention for SFA intake ( in gram). The intake was measured through interview using two replicates 24-hour food recall on non-consecutive days. The foods were converted to energy and nutrients based on Indonesia food composition tables available in nutrisurvey software.
Change in PUFA/SFA (P/S) ratio | baseline (before intervention and end-line (after 12-weeks interventions)
  Change from baseline at 12-week intervention for P/S
Change in dietary fiber intakes | baseline (before intervention and end-line (after 12-weeks interventions)
  Change from baseline at 12-week intervention for dietary fiber intake ( in gram). The intake was measured through interview using two replicates 24-hour food recall on non-consecutive days. The foods were converted to energy and nutrients based on Indonesia food composition tables available in nutrisurvey software.
Change in iron (Fe) intake | baseline (before intervention and end-line (after 12-weeks interventions)
  Change from baseline at 12-week intervention for iron intake ( in mg). The intake was measured through interview using two replicates 24-hour food recall on non-consecutive days. The foods were converted to energy and nutrients based on Indonesia food composition tables available in nutrisurvey software.
Change in zinc (Zn) intake | baseline (before intervention and end-line (after 12-weeks interventions)
  Change from baseline at 12-week intervention for zinc intake ( in mg). The intake was measured through interview using two replicates 24-hour food recall on non-consecutive days. The foods were converted to energy and nutrients based on Indonesia food composition tables available in nutrisurvey software.

SECONDARY OUTCOMES:
Change in Body weight | baseline (before intervention and end-line (after 12-weeks interventions)
  Change in Body weight (in Kg) from baseline at 12-week intervention
Change in waist circumference | baseline (before intervention and end-line (after 12-weeks interventions)
  change of waist circumference (in cm), from baseline at 12-week intervention
Change in total cholesterol level | baseline (before intervention and end-line (after 12-weeks interventions)
  Change of total cholesterol (in mg/dL) from baseline at 12-week intervention
Change in Low Desnsity Lipoprotein (LDL) cholesterol | baseline (before intervention and end-line (after 12-weeks interventions)
  Change of LDL (in mg/dL) from baseline at 12-week intervention
Change in serum High Density Lipoprotein (HDL) cholesterol | baseline (before intervention and end-line (after 12-weeks interventions)
  Change of HDL (mg/dL) from baseline at 12-week intervention
Change in serum triglyceride (TG) | baseline (before intervention and end-line (after 12-weeks interventions)
  Change of TG (mg/dL) from baseline at 12-week intervention

OTHER OUTCOMES:
Change in Body Mass Index | baseline (before intervention and end-line (after 12-weeks interventions)
  Change in body mass index (kg/m2) from baseline at 12-week intervention, calculated from body weight (in kg) divided by square body height (in meter suquare), endline minus baseline
Change in Castelli's Index | baseline (before intervention and end-line (after 12-weeks interventions)
  Change of Castelli's index from baseline at 12-week intervention, calculated from the total cholesterol level divided by serum HDL

CONTACTS AND LOCATIONS:
Overall Officials: Murdani Abdullah, Study Chair — Indonesia University
Locations (1):
- Dinas Kesehatan Kota Padang, Padang, West Sumatra, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gusnedi G, Fahmida U, Witjaksono F, Nurwidya F, Mansyur M, Djuwita R, Dwiriani CM, Abdullah M. Effectiveness of optimized food-based recommendation promotion to improve nutritional status and lipid profiles among Minangkabau women with dyslipidemia: A cluster-randomized trial. BMC Public Health. 2022 Jan 6;22(1):21. doi: 10.1186/s12889-021-12462-5. PMID 34991541